CLINICAL TRIAL: NCT04030819
Title: Effectiveness of a Schema Therapy on Anxiety in Patients With Multiple Sclerosis .a Randomized Control Study in 106Persian Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: Effectiveness of a Schema Therapy on Anxiety in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paris Nanterre University (Other)
Collaborators: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Azam Mansourzadeh, PHD student of university Nanterre-clinical researcher in university ISFAHAN, Paris Nanterre University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ParisNU
Record Dates: First submitted 2019-07-11; First posted 2019-07-24 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Anxiety
Keywords: anxiety; multiple sclerosis; schema therapy
MeSH Terms: conditions — Anxiety Disorders; Multiple Sclerosis | interventions — Schema Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention
- experimental group (Experimental): schema therapy
  Interventions: Behavioral: schema therapy

INTERVENTIONS:
Behavioral: schema therapy — The intervention is the schema therapy focuses on the management of anxiety and is based on self-efficacy, self-management . It consists of 20 once-weekly sessions of 90 minutes (with a 15 Min break), with homework activities between the sessions
  Arms: experimental group

SUMMARY:
It is a multicentric randomized and controlled study comparing a Scheme therapy program versus local practice in RRMS patients with anxiety. Patients will assist to twenty once-weekly group sessions with a 6-month follow up after the end of the programme. The main criteria is the impact of schema therapy on anxiety evaluated by the questionnaires at the end of the program and at the end of the 6-month follow-up.

DETAILED DESCRIPTION:
A parallel arm randomized controlled trial comparing a group receiving Scheme Therapy plus current usual practice versus a group receiving current local practice only. The trial will take place in KASHANI Hospital (in Isfahan).Recruitment of the participants will be identified and recruited by the neurologists of the hospitals who take part in the programme, when they come for a medical examination.

After giving their informed consent, the patients will be entered onto the trial database and randomized to either the schema therapy or control using software allocated The intervention is the schema therapy focuses on the management of anxiety and is based on self-efficacy, self-management . It consists of 20 once-weekly sessions of 90 minutes (with a 15 Min break), with homework activities between the sessions. It is designed for groups of 8 people and will be delivered by two psychologists. The programme is standardized: Power Points presentations support each session and a detailed therapist manual and companion patient workbook accompany the programme.

For the ST group an evaluation will be administered pretest and post-test six months after the end of the schema therapy programme and at the same times for those in the control group. Socio-demographic and medical data, age, sex, level of education, marital status, number of children and professional status; date of diagnosis, disease type, level of disability (EDSS, Kurtzke, 1983) and information on relapses and treatments, are evaluated. The main criteria is the impact of schema therapy on anxiety evaluated by the BAI (beck anxiety inventory ) and level of cortisol at 6 month after the start program . Secondary criteria are: impact on the psychological dimensions assessed by Hospital Anxiety and Depression Scale (HADS), intensity of fatigue assessed by Fatigue Severity Scale (FSS), sleep quality evaluated by the Pittsburgh Sleep Quality Index(PSQI) depression by BDI (beck depression inventory ) and quality of life evaluated by (Multiple sclerosis impact scale) MSIS29.

ELIGIBILITY:
Inclusion Criteria:

* subject has relapsing remitting MS
* anxiety (score >26 at the BAI scale)
* history of psychotic disorders
* history of cognitive deficiency
* use anti-depressant in the past 3 months
* history of relapse in the past 3 month
* expanded Disability Status Scale score less than 6
* ability reading and writing Persian
* Non hospitalized

Exclusion Criteria:

* history of psychotic disorders
* history of cognitive deficiency
* use anti-depressant in the past 3 months
* history of relapse in the past 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
changes Anxiety in patient with MS,Beck Anxiety Inventory (BAI) | Change measures in 0,6,12 month
  Beck Anxiety Inventory (BAI),self-reported questionnaire of anxiety,.21-question multiple- choice each answer being scored on a scale value of 0 (not at all) to 3 (severely),Higher total scores indicate more severe anxiety symptoms . score between 0-63
changes in level of cortisol | Change measures in 0,6,12 month
  cortisol measure by Immunoassay by cortisol saliva ELISA, DiaMetra ( kit),adult morning peak :3-10 ,higher values represent more anxiety

SECONDARY OUTCOMES:
changes in depression,Beck Depression Inventory (BDI) | Change measures in 0,6,12 month
  Beck Depression Inventory (BDI)- self report questionnaires,21-question multiple-choice,each answer being scored on a scale value of 0 (not at all) to 3 (severely),total scores indicate more severe depression symptoms . score between 0-63
changes quality of life.Multiple sclerosis impact scale - 29 items(MSIS29) | Change measures in 0,6,12 month
  Multiple sclerosis impact scale - 29 items.self -reported questionnaires (MSIS29):29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale,Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
changes in quality of sleep.Pittsburgh Sleep Quality Index (PSQI) | Change measures in 0,6,12 month
  Pittsburgh Sleep Quality Index (PSQI) : self-report questionnaire that assesses sleep quality over a 1-month time intervalself-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items,Each item is weighted on a 0-3 interval scale The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality..
changes in fatigue.Fatigue Severity Scale (FSS) | Change measures in 0,6,12 month
  Fatigue Severity Scale (FSS). self -reported questionnaires The FSS questionnaire contains nine statements that attempt to explore severity of fatigue symptoms.each item being scored on a scale value of 1 to 7. score between 9-63.higher the score indicate greater fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Marie claire GAY, full prof, Study Director — university paris Nanterre; vahid shaygannejad, professor, Study Director — Isfahan university of medical science; AZAM Mansourzadeh, Principal Investigator — university paris Nanterre
Locations (1):
- university Paris Nanterre, Paris, France

IPD SHARING:
Plan to Share IPD: No